CLINICAL TRIAL: NCT00327210
Title: Blood Glucose Awareness Training Delivered Over the Internet (BGATHome.Com): Feasibility and Efficacy
Brief Title: Feasibility and Efficacy of Delivering Blood Glucose Awareness Training Over the Internet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11593
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: BGAT; Blood Glucose Awareness Training; Diabetes; T1DM; Internet; Web; Intervention; Treatment; Behavior; Education; Awareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BGATHome (Experimental): Blood Glucose Awareness Training at Home Internet Intervention
  Interventions: Behavioral: Blood Glucose Awareness Training
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Blood Glucose Awareness Training
  Arms: BGATHome

SUMMARY:
BGATHome is an interactive, web-based training program designed to improve the ability of adults with Type 1 Diabetes to recognize, predict, treat, and avoid extreme blood glucose (BG) events. It was developed at the University of Virginia over the past 20 years with funding from the National Institutes of Health and the American Diabetes Association. BGATHome provides important knowledge about personal insulin use, food, and activity regimens that influence BG levels. Users of this program will learn to monitor and recognize the cues that signal hyper and hypoglycemic events, and enhance their ability to control these fluctuations.

DETAILED DESCRIPTION:
Interested subjects will be informed that they will be randomly assigned to either receive the BGATHome program or will be placed in a wait-list control group. Respondents will be informed that if they are in the control group, they are expected to complete the pre- and post-assessments (HHC and questionnaires), but once these are complete, they will be given free access to the BGATHome program. Respondents will be informed that being in the control group will delay their access to the program by approximately 5 months.

A hand held computer (PDA) will be provided for use during this study. Subjects will be asked to first estimate their blood glucose level and enter this estimate into the PDA. They will then actually measure their blood glucose level and enter this actual value into the PDA also. This process of first estimating the blood glucose level and then taking an actual reading will be repeated 70 times during the 4-week period. The time estimated for this task is approximately 3 minutes for entering each estimate and measurement, or a total of 3.5 hours over the 4 weeks. The PDA device will be returned (postage paid) after the first 4 weeks of the study. At 12 weeks, the device will be sent to study subjects again and the process of obtaining data about blood glucose levels by first estimating and then taking an actual reading will be repeated over the next 4 weeks, as before. The PDA device will again be returned (postage paid) after 4 weeks of data collection. The total amount of time estimated to enter data into a PDA for this study is approximately 7 hours.

Subjects will be asked to respond to a series of four questionnaires on the Internet, taking approximately 30-45 minutes. These questionnaires will be completed 3 times over the course of the study - before beginning the BGATHome program, at 12 weeks and at one year after completing the BGATHome program. The total time estimated to complete the three sets of questionnaires is approximately 2 hours, 15 minutes.

Experimental subjects will be asked to complete a total of eight units of the BGATHome program, completing one unit a week except for the first week when two units will be completed. Each unit will take approximately one hour to complete. Subjects will have a maximum of 12 weeks to complete BGATHome. The total time is estimated at 8 hours.

The wait-list control subjects will be offered access to the BGATHome program approximately five months after consenting to be in the study. They will then complete the series of four questionnaires on the Internet 12 weeks after using the BGATHome program. If the control subjects do not choose to use the program, a one year follow assessment will occur like the experimental subjects.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least one year.
* Access to the Internet.
* Routinely perform Self Monitoring of Blood Glucose at least three times a day.
* ≥ 21 years of age

Exclusion Criteria:

- Not able to complete the Internet program in 12 weeks.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Feasibility | 12 weeks
  Internet Evaluation

SECONDARY OUTCOMES:
Improved blood glucose awareness | 12 weeks
  Blood Glucose Diaries
Reduced adverse events | 12 weeks
  Blood Glucose Diaries
Improved psychological functioning | 12 weeks
  Hypo Fear Survey, Diabetes Quality of Life
Improved knowledge | 12 weeks
  Diabetes Knowledge Scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cox, Ph.D, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Viginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Cox D, Ritterband L, Magee J, Clarke W, Gonder-Frederick L. Blood glucose awareness training delivered over the internet. Diabetes Care. 2008 Aug;31(8):1527-8. doi: 10.2337/dc07-1956. Epub 2008 May 13. PMID 18477813